CLINICAL TRIAL: NCT02869412
Title: A Physical Activity Behavior Change Guide for Prostate Cancer Patients (iTRAIN Study)
Brief Title: Computer-Based Behavior Change Guide in Increasing Physical Activity in Patients With Prostate Cancer Who Have Received Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Esther Moe, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00011113; NCI-2016-01217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CPC-14128-L; 11113; IRB00011113 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (BCG website) (Experimental): Patients use the BCG website which will collect personal information including individual health priorities/goals, demographics (i.e. age, ethnicity), health information (i.e. weight, height, cancer history, other health conditions), individual capabilities, physical activity level, and exercise preferences. Patients then receive a report with a personalized physical activity plan.
  Interventions: Other: Computer-Assisted Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (passive website) (Active Comparator): Patients use a passive website (American Cancer Society Guidelines on Nutrition and Physical Activity for Cancer Survivors).
  Interventions: Other: Computer-Assisted Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Computer-Assisted Intervention — Use BCG website
  Arms: Group I (BCG website)
Other: Computer-Assisted Intervention — Use passive website
  Arms: Group II (passive website)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies how well a computer-based behavior change guide works in increasing physical activity in patients with prostate cancer who have received androgen deprivation therapy. A computer-based behavior change guide website may increase physical activity level for prostate cancer survivors and help doctors understand what outcomes related to becoming physically active are most important to patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Engage with prostate cancer patients (PCPs) who have received or are currently on androgen deprivation therapy (ADT) to develop a computer-based behavior change guide (BCG) for PCPs to provide fundamental information about benefits of exercise for their individual capabilities and goals and provide a personalized physical activity plan. (Development Phase) II. Engage with PCPs to understand what outcomes are most important to them related to becoming active (e.g., helped me manage side-effects of treatment, reduced fatigue) and develop measures to evaluate these patient-centered outcomes. (Development Phase) III. Evaluate the BCG in a study comparing the personalized computer-based BCG with physical activity recommendations provided via a passive website (American Cancer Society Guidelines on Nutrition and Physical Activity for Cancer Survivors) among PCPs who have received ADT. (Evaluation Phase)

OUTLINE:

DEVELOPMENT PHASE: Patients view mock-ups of the BCG web design on a computer, iPad, or printed color paper and provide feedback with a one-on-one interview or separately using the think/talk aloud method followed by a one-on-one interview. After completion of these design rounds, patients use the BCG website and provide individual feedback.

EVALUATION PHASE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients use the BCG website which will collect personal information including individual health priorities/goals, demographics (i.e. age, ethnicity), health information (i.e. weight, height, cancer history, other health conditions), individual capabilities, physical activity level, and exercise preferences. Patients then receive a report with a personalized physical activity plan.

GROUP II: Patients use a passive website (American Cancer Society Guidelines on Nutrition and Physical Activity for Cancer Survivors).

After completion of study, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer (PCa) diagnosis
* Able to read English on a computer screen
* Signed an Institutional Review Board (IRB)-approved informed consent
* EVALUATION PHASE
* Underactive (defined as physically active for less than 30 minutes per day fewer than 2 days per week)
* Access to a computer at home or public location

Exclusion Criteria:

* Non-English speaking subjects are excluded from this study; the website being developed will only be available in English

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in self efficacy for exercise, assessed by the Self Efficacy for Exercise questionnaire (Evaluation Phase) | Baseline up to 2 months
  For the qualitative characteristics collected, univariate summaries (e.g., frequency counts and proportions) will be calculated. For quantitative characteristics, means, standard deviations, medians, and ranges will be computed. The analysis will be conducted as an intent-to-treat efficacy assessment comparing the two interventions. Analyses will examine changes between baseline and follow-up scores on outcome measures by group. Comparisons will be conducted using Generalized Estimating Equations (GEE) with robust (sandwich) variance estimates.
Stage of change for exercise, assessed by the Stage of Change for Exercise questionnaire (Evaluation Phase) | Up to 2 months
  For the qualitative characteristics collected, univariate summaries (e.g., frequency counts and proportions) will be calculated. For quantitative characteristics, means, standard deviations, medians, and ranges will be computed. The analysis will be conducted as an intent-to-treat efficacy assessment comparing the two interventions. Analyses will examine changes between baseline and follow-up scores on outcome measures by group. Comparisons will be conducted using GEE with robust (sandwich) variance estimates.
Website usability, assessed by qualitative evaluation of interviews and feedback (Development Phase) | Up to 9 months

SECONDARY OUTCOMES:
Average activity level for seniors per Community Healthy Activity Model Program for Seniors (CHAMPS) questionnaire | Baseline up to 2 months
  CHAMPS is a 41-item questionnaire developed by UCSF that asks about recent participation in specific physical activities and structured exercise to measure changes in physical activity level in older adults (age 65 and up). This questionnaire estimates total weekly energy expenditure (in kilocalories per week) from low to vigorous intensity physical activities for older adults. This physical activity survey has been used and validated with cancer survivors. The 41-item questionnaire asks about engagement in vigorous, moderate, and light activities per week, including frequency and duration, du
Body weight | Baseline up to 2 months
  Participants will be asked to self-report their current weight in pounds.
Measurement of exercise motivation using the Behavioral Regulation In Exercise Questionnaire (BREQ) | Baseline up to 2 months
  This questionnaire concerns the reasons why a person exercises regularly, works out, or engages in other such physical activities. It is structured so that it asks one questions and provides responses that represent external regulation, introjected regulation, identified regulation, and intrinsic motivation. The basic issue concerns the degree to which one feels autonomous with respect to exercising or engaging in physical activity. The BREQ measures the continuum of behavioral regulation in exercise psychology research. The original BREQ (Mullan, Markland & Ingledew, 1997) was developed to me
Measurement of fatigue using the Piper Fatigue Scale | Baseline up to 2 months
  The Piper Fatigue Scale measures fatigue in cancer research, and includes subdomains of behavioral, affective, sensory, and cognitive/mood attributes of fatigue. The Piper Fatigue Scale-12 is an instrument to measure the subjective dimension of fatigue, developed by BF Piper, AM Lindsey, MJ Dodd, S Ferketich, SM Paul and S Weller. The Piper Fatigue Scale is one of the commonly used multidimensional fatigue measures in the cancer research field and includes subdomains of behavioral, affective, sensory, and cognitive/mood attributes of fatigue.
Measurement of quality of life per European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire-core 30 (QLQ-C30) questionnaire | Baseline up to 2 months
  EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The QLQ-C30 incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. Scores range from 0-100, with higher functional scale scores indicating a higher level of healthy fu
Self-reported physical activity assessed by the Rapid Assessment of Physical Activity (RAPA) | Baseline up to 2 months
  The RAPA questionnaire was designed to provide clinicians with a tool for quickly assessing the level of physical activity of their older adult patients. It was developed after a review and evaluation of existing written questionnaires. The RAPA questionnaire was developed by University of Washington Health Promotion Research Center to provide clinicians with a tool for quickly assessing the level of physical activity of their older adult patients.
Website use and acceptability assessed by questionnaire | Responses collected at 2 months
  Questions about participant use and their perception of the website's features and usability will provide insights into the acceptability to revise it for further development. This is a study specific questionnaire developed to measure the frequency of use of the websites and participant preferences about exercise. Higher scores indicate better use and acceptance of the exercise information and website. In addition, the questionnaire includes an open ended question for participants to provide the study team with any additional thoughts or comments about the website.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Moe, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States